CLINICAL TRIAL: NCT03806140
Title: Proof-of-Concept of an Infrastructure for Text Messaging Interventions at CHOP: Development and Evaluation of THRIVE (Texting Health Resources to Inform, motiVate, and Engage)
Brief Title: Development and Evaluation of THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-010834
Record Dates: First submitted 2019-01-10; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Oncology
Keywords: Texting; mHealth; Adolescents and young adults transitioning of treatment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Receive daily text messages
  Interventions: Behavioral: text messages
- Control group (No Intervention): No text messages, only written educational materials

INTERVENTIONS:
Behavioral: text messages — receive about one health-related text message a day for 16 weeks
  Arms: Intervention group

SUMMARY:
Investigators will test the feasibility and acceptability, as well as efficacy (exploratory aim) of a text messaging intervention for Adolescents and young adults (AYA) transitioning off active treatment for cancer. Texting Health Resources to Inform, motiVate, and Engage (THRIVE) is intended to improve knowledge about health promotion and health vulnerability and importance of continued engagement in care, while also providing support and improving efficacy to achieve health-related goals.

DETAILED DESCRIPTION:
Adolescents and young adults (AYA) with cancer are recognized as an understudied and underserved population in oncology. AYA engagement in ongoing disease management is compromised by lack of awareness of their continued health vulnerabilities and need for continued care, their desire to be "normal" and remove themselves from the cancer experience, and lack of AYA-appropriate support and services. Thus, AYA with cancer, especially those completing active treatment, are extremely vulnerable and in need of support to maintain remission and assure optimal health into adulthood. To address the immediate need for innovative interventions targeting AYA completing cancer treatment, the proposed study will test the efficacy, feasibility, and acceptability of a tailored text messaging intervention for AYA transitioning off active treatment called THRIVE (Texting Health Resources to Inform, motiVate, and Engage).

A pilot randomized controlled trial testing the acceptability and feasibility (primary) and initial efficacy (secondary) of a health promoting mobile health texting intervention with AYA transitioning off active cancer treatment to follow-up care.

The intervention compares a texting intervention to a receipt of an AYA survivorship handbook. Acceptability and feasibility are primary outcomes. Efficacy outcomes include measures of knowledge, healthcare utilization, adherence, engagement in care, and psychosocial well-being measures.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with cancer
2. Males or females between the ages of 12 and 25
3. In remission (per documentation in chart)
4. Within 12 months of completing active treatment for cancer
5. Cognitively capable to complete measures (per documentation in chart of impairment or parent or provider report).
6. Able to read and speak English.
7. Parent available to provide consent for those ages 12 to 17

Exclusion Criteria:

1)Subjects that do not meet inclusion criteria described above will be excluded.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of promoting a tailored text messaging intervention for AYA transitioning off active treatment | 16 weeks
  All patients will complete a measure of acceptability at the outcome data collection-. The questionnaire consists of 27 items for the control group and 31 items for the intervention group. Items will be answered on a Likert-scale and one open-ended question intended to elicit suggestions for improving the intervention. Items pertain to perceived value, appropriateness, convenience and helpfulness of the intervention.
Number of patients completed 16 week measures | 16 weeks
  Completion of follow-up measures which will be logged by research team for feasibility
Number of patient-reported barriers to technology of text messages | 16 weeks
  Number of participants who report barriers or issues with the text messages and technology for feasibility

SECONDARY OUTCOMES:
Health competence beliefs | 16 weeks
  Health Competence Beliefs Inventory (HBCI) survey - The HCBI assess beliefs about the psychological and functional impact of past medical issues, perceived competence to manage current and future medical issues, perceived medical vulnerability now and in the future, and perceived connection to/communication with others about medical issues. HCBI includes 4 subscales (autonomy, health vulnerability, cognitive competence, and satisfaction with health care). For this study, we are omitting the cognitive competence subscale, resulting in 16 items.
Engagement in health promoting behaviors | 16 weeks
  Engagement in health promoting behaviors will be assessed using the Health Behavior Survey (HBS). This measure is composed of the 30-item Health Behavior Survey (HBS) that was developed for a previous study (Hocking, Schwartz, Hobbie et al., 2013). HBS alcoholic beverage consumption (4-items), smoking (2-items), other drug use (4-items), sunscreen use (1-item), health-screening (1-item), exercise (4-items), sexual behavior (3-items), and nutrition/weight (7-items). These items will be scored as either health promoting or health limiting (1 point for each health promoting behavior). The total score, as well as scores from each content area, will be used.
Changes in health competence beliefs | 16 weeks
  Perceived Health Competence Scale (PHCS) survey will be used to assess health competence beliefs. The survey is an 8-item instrument designed to assess perceived effectiveness carrying out health behaviors and influencing personal health outcomes. Participants rate each item on a 5-point Likert scale, from strongly disagree to strongly agree. Items yield a total score.
Changes in health related quality of life (HRQL) in adolescent and young adult survivors of childhood cancer | 16 weeks
  Minneapolis-Manchester Quality of Life Instrument-adolescent (MMQL) survey will be used to measure health related quality of life in adolescent and young adult survivors of childhood cancer by assessing physical functioning, psychological functioning, social functioning, cognitive functioning, body image, outlook on life, and intimate relationships. Scores range from one to five, with a higher score indicating a better HRQL An overall QoL score is reached by finding the mean score for all the items.
Patient adherence to clinic attendance | 16 weeks
  Medical record review as well as completion of the Medical Adherence Measure (MAM) survey will be used to assess patient adherence to clinic attendance. The MAM assesses adherence. Patient adherence to medication and to clinic attendance are each rated on a 10-point scale (1 = never; 10 = always take medication). Participants also select barriers to adherence from a list of 12 and the option to write in another reason.
Knowledge of health promoting behaviors | 16 weeks
  Knowledge of health promoting behaviors will be assessed using the Knowledge Acquisition Measure questionnaire. The measure was developed by the research team for use in this study. The questionnaire consists of 23 multiple choice items regarding knowledge of basic health-promoting behaviors (e.g. recommended sunscreen use and maintenance of physical health) as well as five goal-specific questions that each participant will answer based on the goal he or she chose at the time of enrollment. All components of the Knowledge Acquisition Measure aim to assess the amount of health-related knowledge gained over the course of the intervention.
Changes in sleep quality | 16 weeks
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQUI) questionnaire- 19-item self-report questionnaire that measures subjective sleep quality and disturbance in adults over the past one-month period and discriminates "good" and "poor" sleepers (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989). The PSQI yields a global score (PSQI-G) and seven subscale scores consisting of Sleep Quality, Sleep Latency, Sleep Duration, Sleep Efficiency, Sleep Disturbances, Sleep Medications, and Daytime Dysfunction, with a global score of > 5 thought to be suggestive of significant sleep disturbance.
Medication adherence | 16 weeks
  Medical adherence will be assessed by medical record review as well as Medical Adherence Measure (MAM) - Patient adherence to medication and to clinic attendance are each rated on a 10-point scale (1 = never; 10 = always take medication). Participants also select barriers to adherence from a list of 12 and the option to write in another reason.
Fatigue | 16 weeks
  Multidimensional fatigues scale (MFS) questionnaire will be used to assess fatigue. The measure is an 18- item questionnaire that yields a total score and three subscale scores: General Fatigue, Sleep/Rest Fatigue, and Cognitive Fatigue. Items are answered on a 5-point Likert-type scale indicating how problematic each element of fatigue was over the past month. Lower scores indicate more fatigue
Attainment of health related goals | week 1 and 16
  Goal Attainment Measure - was developed for this study, and assesses participants' expectation of (10-items) and progress related to achieving their chosen goal (9-items).
Patient adherence to medication compliance | 26 weeks
  medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Schwartz, PhD, Principal Investigator — Children's Hospital of Philadelphia

IPD SHARING:
Plan to Share IPD: No